CLINICAL TRIAL: NCT01357863
Title: Clinical Outcomes on ErbB2+ MBC Patients Treated With Lapatinib-Capecitabine After Trastuzumab Progression: Role of Early Versus Late Switch to Lapatinib-Capecitabine (TYCO1) - Brazil
Brief Title: Role of Early Versus Late Switch to Lapatinib-Capecitabine
Acronym: (TYCO1)
Status: Terminated | Type: Observational
Why Stopped: This study was terminated because the National Ethics Committee has not approved the protocol.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 113960
Record Dates: First submitted 2011-05-19; First posted 2011-05-23 (Estimated); Last update posted 2018-09-14 (Actual); Status verified 2018-05

CONDITIONS: Cancer
Keywords: Lapatinib; Observational Study; Trastuzumab; Brazil; Metastatic Breast Cancer
MeSH Terms: conditions — Neoplasms; Breast Neoplasms | interventions — Therapeutics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients on second line treatment: Patients treated with Lapatinib-capecitabine immediately after first Trastuzumab-containing regimen progression
  Interventions: Drug: Treatment
- Patients on third or more lines treatment: Patients treated with Lapatinib-capecitabine after 2 or more lines of treatment after first Trastuzumab-containing regimen progression
  Interventions: Drug: Treatment

INTERVENTIONS:
Drug: Treatment — Patients treated with Lapatinib-capecitabine after Trastuzumab progression

SUMMARY:
The study will be conducted as a multicenter prospective observational cohort study, trying to cover almost all Brazilian States, in a population of ErbB2 positive metastatic breast cancer patients, whose disease has progressed after trastuzumab-containing regimen, comparing outcomes in two groups: Group 1: patients receiving Lapatinib-capecitabine immediately after 1st Trastuzumab progression (second line treatment), and Group 2: patients receiving Lapatinib-capecitabine after 2 or more lines of treatment after 1st trastuzumab progression (third line or greater).

DETAILED DESCRIPTION:
All cases of ErbB2 positive metastatic breast cancer, receiving approved standard treatment with lapatinib-capecitabine, after trastuzumab-containing regimen progression in community setting can participate in this observational study, for a period of 12 months of observation since the start of the lapatinib-capecitabine treatment.

ELIGIBILITY:
* Women with ErbB2+ MBC (ErbB2 expression confirmed by immunohistochemistry or FISH/CISH, either in the primary tumor or in the metastasis, according to the institution's common practice);
* Older than 18 years old;
* Have received prior treatment with trastuzumab-containing regimen for ErbB2+ breast cancer;
* Progressing after trastuzumab-containing regimen either used for the treatment of metastatic disease or progressing after adjuvant /neoadjuvant trastuzumab treatment;
* Eligible to start standard treatment with Lapatinib-capecitabine at conventional doses, in the community setting;
* Signed consent to participate and release information for this study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All cases of ErbB2 positive metastatic breast cancer, receiving approved standard treatment with lapatinib-capecitabine, after trastuzumab-containing regimen progression in community setting can participate in this observational study, for a period of 12 months of observation since the start of the lapatinib-capecitabine treatment.
  Centers from private and public settings, which have incorporated Lapatinib treatment in their routine clinical practice, will be included in this study. Data on the country, type of center, and facility name will be collected on the case report form for use in the data analysis.
Sampling Method: Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2010-07-15; Primary Completion 2010-12-13 (Actual); Study Completion 2010-12-13 (Actual)

PRIMARY OUTCOMES:
Time to disease progression (TTP) | One year
  Time from the date of start of Lapatinib-capecitabine treatment until date of documented disease progression by the treating physician, determined by clinical and/or radiological assessment

SECONDARY OUTCOMES:
Overall response rate (ORR) determined by treating physician | One year
  Percentage of patients showing complete response (CR) and partial response (PR) to the given treatment
One year overall survival (OS) | One year
  Time from the start of lapatinib-capecitabine treatment until death due to any cause (measured at the end of follow-up)
Serious adverse events (SAEs) | One year
  Describe lapatinib-related spontaneous reported serious adverse events
Clinical Global Impression (CGI) | One year
  CGI assessment by the treating physician in the last visit (visit 4 or discontinuation visit)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (10):
- Brazil (10):
  - GSK Investigational Site, Vitória, Espírto Santo
  - GSK Investigational Site, Salvador, Estado de Bahia
  - GSK Investigational Site, Goiânia, Goiás
  - GSK Investigational Site, Natal, Rio Grande do Norte
  - GSK Investigational Site, Porto Alegre, Rio Grande do Sul
  - GSK Investigational Site, Florianópolis, Santa Catarina
  - GSK Investigational Site, São José dos Campos, São Paulo
  - GSK Investigational Site, Belo Horizonte
  - GSK Investigational Site, Rio de Janeiro
  - GSK Investigational Site, São Paulo